CLINICAL TRIAL: NCT01670539
Title: PILOT: Home Telemonitoring for Self-Management Education of Patients With Lung Ca
Brief Title: Home Telemonitoring for Patients With Lung Cancer
Acronym: HTPLC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-22930; 1R15CA150999 (NIH)
Record Dates: First submitted 2012-08-09; First posted 2012-08-22 (Estimated); Results first posted 2022-01-20 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2021-12

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Telemonitoring; Rural; Nursing
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telemonitor (Experimental): In addition to routine care, the "HomMed Telemonitor" wireless telemonitoring system (intervention)will be used in the patient's home for 14 days to alert the clinical research nurse to changes in patients conditions in order to contact them to teach self-management. The Honeywell HomMed Genesis™ DM Remote Patient Care Monitor will be used to measure temperature, pulse, oxygen level,weight and blood pressure. The telemonitor will also ask for a YES or NO response to questions on symptoms such as difficulty breathing. Research nurses review the data daily and call the participant for 2 weeks, and continue to monitor outcomes for 2 months.
  Interventions: Device: HomMed Telemonitor
- Routine care for patients with lungCa (No Intervention): Traditional physician ordered post-hospital care for patients with lung CA in rural WV requires patients to make an outpatient office/ clinic visit two to three weeks after discharge;a few patients receive homecare service referrals. No attempt to change care - just monitor what is used and collect study data at Discharge, 2 weeks, one month and two months.

INTERVENTIONS:
Device: HomMed Telemonitor — A "HomMed Telemonitor" wireless telemonitoring system collects data on a daily basis, including heart rate, blood pressure, oxygen level, body temperature, weight, responses to 9 pre-programmed questions (including difficulty breathing, fatigue, limited activities, difficulty taking meds, pain). Telemonitored results are transmitted to the research office for analysis and contact to patient by clinical research nurses.
  Other Names: Honeywell HomMed Genesis™ DM Remote Patient Care Monitor; http://hommed.com/Products/Genesis_DM.asp
  Arms: Telemonitor

SUMMARY:
The purpose of this study is to learn more about using a home machine "Telemonitor" to find problems people with lung cancer may have after being discharged from the hospital and help them manage problems by contacting their healthcare provider.The study hypothesis is that patients with lung CA using short-term (14 days)home telemonitors, educated/coached by nurses on telemonitor data risks/implications for the first two weeks after hospital discharge, will be able to self-report their signs/ symptoms to the clinician resulting in decreased use of costly health care resources over 60 days.

DETAILED DESCRIPTION:
All patients in the study will receive usual care after hospital discharge. This study also involves an interview and review of your medical records, and uses the "telemonitor" machine to measure your temperature, pulse, oxygen level,weight and blood pressure. The telemonitor will also ask you to press YES or NO buttons in response to questions on your symptoms such as difficulty breathing. Research nurses will come to your home 3 times and it will take about 30 minutes for each visit for the nurse to record the information using the telemonitor. You will also be asked to fill out a survey about your ability to do activities and your health status. This will take approximately another 30 minutes. You may or may not receive the small telemonitor (about as big as a large book) for 14 days after discharge to provide additional information to the researchers. If you receive the monitor for the full 14 days, you or someone you ask us to train will be taught to use the monitor every morning to collect information on how you will "talk" to you to tell you to put a blood pressure cuff on your arm and an oxygen measurer on your finger. You will step on a scale to take your weight and you will use a forehead sensor to take your temperature. The blood pressure, weight, temperature, your pulse, and your oxygen level will be recorded by the monitor. It will then ask you at least 10 questions and you will push a yes or no button indicating how much difficulty you are having with your daily activities and shortness of breath. The monitor will then connect to your telephone line using a no-charge "800" number and transmit the information to the researchers. If you do not have a phone, a special antenna will be connected to the monitor to transmit the information wirelessly. The nurse will call you every day for the 14 days when you have the monitor. If you do not receive the monitor for the full 14 days, you will still have the monitor used by the nurse when you are visited at least 3 times at home to gather information on how you are doing after hospital discharge. These home monitor visits will be within 2 days after discharge, 2 weeks after discharge, and 2 months after discharge. The main difference is that the monitor will not be left in your home but will be brought by the nurse on each visit. You will also receive a phone call to ask you questions about the study at 1 month after discharge. If you do not have a phone, you will receive another home visit. Whether or not you get the monitor for the full 14 days will be determined randomly by computer before the nurse visits you at home the first time. are doing. The monitor will turn on each day at the same time; the monitor

ELIGIBILITY:
Inclusion Criteria:

(1) patients admitted to the hospital for lung CA as a primary or secondary diagnosis; (2) at least 45 years of age and up to 90 years old; (3) stable mental status and ability to speak (but not necessarily read) the primary language of the region (English).

Exclusion Criteria:

1. are not discharged to home settings
2. are discharged to hospice
3. display a verbalized inability to understand or answer the questionnaires, (4) are disqualified at the discretion of the treating physician, and/or (4) live beyond a 75 mile radius of the hospital.

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Georgia L Narsavage, PhD, MSN, Principal Investigator — West Virginia University
Locations (1):
- WVU Mary Babb Randolph Cancer Center and Ruby Hospital, Morgantown, West Virginia, United States

REFERENCES:
- [Background] Chen YJ, Narsavage GL, Culp SL, Weaver TE. The development and psychometric analysis of the short-form Pulmonary Functional Status Scale (PFSS-11). Res Nurs Health. 2010 Dec;33(6):477-85. doi: 10.1002/nur.20403. Epub 2010 Oct 18. PMID 20957666
- [Background] Narsavage G, Romeo E. Education and support needs of younger and older cancer survivors. Appl Nurs Res. 2003 May;16(2):103-9. doi: 10.1016/s0897-1897(03)00008-9. PMID 12764721
- [Background] Narsavage GL, Naylor MD. Factors associated with referral of elderly individuals with cardiac and pulmonary disorders for home care services following hospital discharge. J Gerontol Nurs. 2000 May;26(5):14-20. doi: 10.3928/0098-9134-20000501-08. PMID 11111516

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from West Virginia University Ruby Memorial Hospital (WVUH) and the Mary Babb Randolph Cancer Center (MBRCC) at WVUH. The study subject recruitment began in April, 2011 and terminated at the end of December 2012.
Pre-assignment Details: Two visits were needed in hospital to explain study prior to requesting consent in order to address literacy and provide opportunity for family member to be present. Time 1 data were collected at time of consent and then patients were assigned to groups prior to discharge.
Groups:
- Telemonitor: In addition to routine care, the "HomMed Telemonitor" wireless telemonitoring system (intervention)will be used in the patient's home for 14 days to alert the clinical research nurse to changes in patients conditions in order to contact them to teach self-management. The Honeywell HomMed Genesis™ DM Remote Patient Care Monitor will be used to measure temperature, pulse, oxygen level,weight and blood pressure. The telemonitor will also ask for a YES or NO response to questions on symptoms such as difficulty breathing. Research nurses review the data daily and call the participant for 2 weeks, and continue to monitor outcomes for 2 months.
  HomMed Telemonitor: A "HomMed Telemonitor" wireless telemonitoring system collects data on a daily basis, including heart rate, blood pressure, oxygen level, body temperature, weight, responses to 9 pre-programmed questions (including difficulty breathing, fatigue, limited activities, difficulty taking meds, pain).
Period: Overall Study
Arm/Group | Telemonitor | Routine Care for Patients With lungCa
Started | 26 | 21
Completed | 20 | 16
Not Completed | 6 | 5
Not completed — Death | 3 | 5
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Population: PI has left the institution and a report about the results was found, but the information within the report is not always broken down between the arms.
Groups:
- Telemonitor and Routine Care for Patients With lungCa: PI left the institution and demographic information was not broken down into arms.
  Telemonitor:
  In addition to routine care, the "HomMed Telemonitor" wireless telemonitoring system (intervention)will be used in the patient's home for 14 days to alert the clinical research nurse to changes in patients conditions in order to contact them to teach self-management. The Honeywell HomMed Genesis™ DM Remote Patient Care Monitor will be used to measure temperature, pulse, oxygen level,weight and blood pressure. The telemonitor will also ask for a YES or NO response to questions on symptoms such as difficulty breathing. Research nurses review the data daily and call the participant for 2 weeks, and continue to monitor outcomes for 2 months.
  HomMed Telemonitor: A "HomMed Telemonitor" wireless telemonitoring system collects data on a daily basis, including heart rate, blood pressure, oxygen level, body temperature, weight, responses to 9 pre-programmed questions (including difficulty breathing, fatigue, limited activities, difficulty taking meds, pain).
  Routine care for patients with lungCa:
  Traditional physician ordered post-hospital care for patients with lung CA in rural WV requires patients to make an outpatient office/ clinic visit two to three weeks after discharge;a few patients receive homecare service referrals. No attempt to change care - just monitor what is used and collect study data at Discharge, 2 weeks, one month and two months.
Arm/Group | Telemonitor and Routine Care for Patients With lungCa
Number analyzed (Participants) | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants] — All efforts have been made to contact the PI, but the only available information is a small results document. The results information found was not always broken down by arm and the gender and race information provided include information from a 10 person sub-study. It cannot be determined which participants were from the sub-study, so information related to gender and race for this specific study cannot be determined. Population: All efforts have been made to contact the PI, but the only available information is a small results document. The results information found was not always broken down by arm and the gender and race information provided include information from a 10 person sub-study. It cannot be determined which participants were from the sub-study, so information related to gender and race for this specific study cannot be determined.
Race (NIH/OMB) [Count of Participants; unit: Participants] — All efforts have been made to contact the PI, but the only available information is a small results document. The results information found was not always broken down by arm and the gender and race information provided include information from a 10 person sub-study. It cannot be determined which participants were from the sub-study, so information related to gender and race for this specific study cannot be determined.
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 0
    More than one race | 0
    Unknown or Not Reported | 47

OUTCOME MEASURES:

1. Primary Outcome: Changes in Telemonitor Data From Baseline: Temperature
Description: Changes in temperature measured by telemonitor daily over 14 days after hospital discharge
Time Frame: 14 days
Population: Results information was not available broken down by arm.
Measure: Mean (Full Range); unit: Degrees Fahrenheit
Arm/Group | Telemonitor and Routine Care for Patients With lungCa
Number analyzed (Participants) | 47
Degrees Fahrenheit | 97.05 [96.6 to 97.5]

2. Primary Outcome: Changes in Telemonitor Data From Baseline: Pulse Rate
Description: Changes in pulse rate measured by telemonitor daily over 14 days after hospital discharge
Time Frame: 14 days
Population: Results information was not available broken down by arm
Measure: Mean (Full Range); unit: beats per minutes (bpm)
Arm/Group | Telemonitor and Routine Care for Patients With lungCa
Number analyzed (Participants) | 47
beats per minutes (bpm) | 93 [89 to 97]

3. Primary Outcome: Changes in Telemonitor Data From Baseline: Blood Pressure
Description: Changes in blood pressure measured by telemonitor daily over 14 days after hospital discharge
Time Frame: 14 days
Population: Results information was not available broken down by arm
Measure: Mean (Full Range); unit: mmHg
Arm/Group | Telemonitor and Routine Care for Patients With lungCa
Number analyzed (Participants) | 47
mmHg
  Diastolic | 69.5 [66 to 73]
  Systolic | 122 [115 to 129]

4. Primary Outcome: Changes in Telemonitor Data From Baseline: SpO2
Description: Changes in SpO2 measured by telemonitor daily over 14 days after hospital discharge
Time Frame: 14 days
Population: Results information was not available broken down by arm.
Measure: Mean (Full Range); unit: percentage of oxygen
Arm/Group | Telemonitor and Routine Care for Patients With lungCa
Number analyzed (Participants) | 47
percentage of oxygen | 93.5 [92 to 95]

5. Primary Outcome: Changes in Telemonitor Data From Baseline: Weight
Description: Changes in weight measured by telemonitor daily over 14 days after hospital discharge
Time Frame: 14 days
Population: Results information was not available broken down by arm.
Measure: Mean (Full Range); unit: pounds
Arm/Group | Telemonitor and Routine Care for Patients With lungCa
Number analyzed (Participants) | 47
pounds | 161.5 [155 to 168]

6. Secondary Outcome: Changes in Telemonitor Symptoms Recorded From Baseline: Dyspnea
Description: Numeric rating for dyspnea, from 0 to 10 with a lower number being a decrease in dysnea. Symptom data requiring yes-no answers to whether the symptom is worse today than yesterday : dyspnea are collected daily via telemonitor for 14 days.
Time Frame: 14 days
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Telemonitor | Routine Care for Patients With lungCa
Number analyzed (Participants) | 26 | 21
score on a scale | 3.8 [3.7 to 3.8] | 2 [2 to 3.1]

7. Secondary Outcome: Changes in Telemonitor Symptoms Recorded From Baseline: Functioning
Description: Pulmonary Functional Status Scale (PFSS-11) , scoring from 0 to 10 with increasing scores indicating an improvement in functioning. Symptom data requiring yes-no answers to whether the symptom is worse today than yesterday : general functioning activities, are collected daily via telemonitor for 14 days.
Time Frame: 14 days
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Telemonitor | Routine Care for Patients With lungCa
Number analyzed (Participants) | 26 | 21
score on a scale | 3.6 [2.8 to 3.6] | 3.2 [3.1 to 3.2]

8. Secondary Outcome: Changes in Telemonitor Symptoms Recorded From Baseline: Pain
Description: Numeric rating for pain (0 to 10 scale) with a lower number indicating less pain. Symptom data requiring yes-no answers to whether the symptom is worse today than yesterday : pain are collected daily via telemonitor for 14 days.
Time Frame: 14 days
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Telemonitor | Routine Care for Patients With lungCa
Number analyzed (Participants) | 26 | 21
score on a scale | 2.8 [2.8 to 4] | 2.8 [2.8 to 3]

ADVERSE EVENTS:
Description: The PI left the institution and a small results document has been found, the documents does not contain adverse events information. All efforts were to made to retrieve adverse events information, but were unsuccessful.
Arm/Group | Telemonitor | Routine Care for Patients With lungCa
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No